CLINICAL TRIAL: NCT03307421
Title: Comparison Between a Team Debriefing With an Instructor and a Team Debriefing Without an Instructor, on Improving Non-technical Skills (TEAM Score) After Simulating a Vital Emergency in a Multidisciplinary Team as Part of the Initial Training
Brief Title: Team Debriefing With Instructor vs Team Debriefing Without Instructor After Simulating a Vital Emergency in a Multidisciplinary Team
Acronym: DEBRIEF-SIM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: ALOUANE Mael (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DEBRIEF-SIM II
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: High Fidelity Simulation Training; Simulation Training
Keywords: simulation; debriefing; team score; multidisciplinarity; DEBRIEF sim II

STUDY DESIGN:
Intervention Model Description: 2 parallel groups, stratified by center, randomized by center
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- debriefing without instructor (Other): Team debriefing without an instructor will be organized as follows. The pairs of participants will be placed in a room with direct access to the video recording of their passage on the simulator. Two documents will be made available to help participants structure their debriefing: one targeting non-technical skills, based on the TEAM Score, and one recalling recommendations on ACR care. Despite its absence at the time of the debriefing, the instructor will be present during the briefing and during the simulation.
  Interventions: Other: debriefing without instructor
- debriefing with instructor (Other): The team debriefing with an instructor will begin immediately after the simulator run and will be governed by the principle of "no judgment" described by Rudolph .
  A portion of the video of the participants' pass may be reviewed and used to support the debriefing (depending on the utility judged by the debrief). Each center will use its own team of trainers, but it will have a predefined plan and predefined objectives, which are provided in advance in order to obtain a standardized debriefing. Moreover, these trainers will not be beginners but will have some expertise in the pedagogy of simulation. They will have to have a DU in a simulation or pedagogy trainer (recommendations from SofraSim) and will have to carry out 15 debriefings per year
  Interventions: Other: debriefing with instructor

INTERVENTIONS:
Other: debriefing without instructor — The randomization will focus on the allocation of the debriefing method: group without instructor versus group with instructor (AI). It will be stratified by center and performed before the first simulation session. The randomization will be carried out by the clinical methodology center of the Besançon University Hospital.
  The sequence of scenarios for each binomial will also be determined by randomization.
  Other Names: video assisted
  Arms: debriefing without instructor
Other: debriefing with instructor — The randomization will focus on the allocation of the debriefing method: group without instructor versus group with instructor (AI). It will be stratified by center and performed before the first simulation session. The randomization will be carried out by the clinical methodology center of the Besançon University Hospital.
  Arms: debriefing with instructor

SUMMARY:
Comparison between a team debriefing with an instructor and a team debriefing without an instructor, on improving non-technical skills (TEAM score) after simulating a vital emergency in a multidisciplinary team as part of the initial training

DETAILED DESCRIPTION:
In spite of the enthusiasm that the simulation raises, its use remains rather complicated in the training of the interns in anesthesiologists-resuscitators (DESAR) and nursing anesthesiologists (EIADE) . Its development has two main limitations: financial and human. Indeed, it mobilizes the medical and paramedical staff already in place, which is a difficulty in a context of demographic constraints.

A simulation session typically takes place in 3 stages: briefing, simulation and debriefing.

The debriefing, the pedagogical pillar of the sessions, demonstrated its influence on the improvement of participants' performances. Different works have tried to define the ideal debriefing method , but its modalities are yet to be defined. To reduce this time Boet and al proposed the assisted video debriefing without instructor. Its principle is that the team of learners will debrief themselves, watching the video recording of their performance. Learners have as a teaching aid a grid that recalls the principles of team work and the technical recommendations of the pathology addressed. This debriefing would therefore reduce the training time and facilitate access to the simulation. However, its pedagogical effectiveness has not been compared to the "gold standard" instructor-team debriefing on initial training and long-term acquisition. The objective of this study is therefore to demonstrate the non-inferiority of a method of debriefing without an instructor (SI) compared to a method of debriefing of team with instructor (AI) on the improvement of a score of non-technical competence (TEAM score) after simulation of a vital emergency in a multidisciplinary team as part of the initial training.

All the DESAR (except the 1st years) and EIADE of the participating centers are eligible. After information on the study and collection of their written consent, the binomials (DESAR + EIADE) will be constituted by drawing lots and randomized by stratification by center, either in debriefing AI or SI.

At D1, they will have a first simulation followed by a debriefing (AI or SI) according to their randomization and immediately after this debriefing, a second simulation. There will be no systematic debriefing behind this second session, but a team of trainers will be able to debrief the binomials that wish to do so. Six months later, the last simulation will take place, followed for all the pairs of an AI debriefing.

The pairs will be evaluated a posteriori, blinded by trained evaluators, for the 3 sessions on a non-technical competence score the TEAM Score and a technical skill score specialized in the pathology encountered. Finally learners will give their self-efficacy before and after each debriefing, and before the 3rd session.

Throughout the course of the study psychological care will be provided: a clearly identified person who is specialized in this pedagogical technique will be present and each participant will have his / her telephone contact details and the usual structures during a psychological distress.

ELIGIBILITY:
Inclusion Criteria:

Common Inclusion Criteria

* Men and women of full age (> 18 years)
* Informed consent signed
* Affiliation to or a beneficiary of a French social security scheme.

Physician Inclusion Criteria

* Internal from 3rd to 10th semester anesthesia resuscitation of the CHU of Besançon, Dijon, Lyon or Strasbourg.

Inclusion Criteria IADE

* IADE students from the nursing school of Besançon, Dijon Lyon or Strasbourg.

Exclusion Criteria:

* Subject without health insurance
* Pregnant woman
* Subject being in the exclusion period of another study or planned by the "National Volunteer File".
* Subject refusing to sign the confidentiality clause
* Internal first-year anesthesia-resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-12-12 (Estimated); Study Completion 2018-12-12 (Estimated)

PRIMARY OUTCOMES:
TEAM SCORE | 6 months
  TEAM Score is a non-technical skills assessment score. This score consists of four items (leadership, teamwork, task management, overall score). Each of these items is rated from 0 to 4, which is a score of 44, to which is added an overall score of 10 points. This score is validated and reflects teamwork skills [30] [31] [32] [33].
  The scoring of the TEAM score will be carried out by a pair composed of a doctor in anesthesia-resuscitation and a nurse anesthetist trained and trained beforehand. This notation will be done afterwards simulations thanks to the registration of passage of the binomials on simulators.

SECONDARY OUTCOMES:
technical score | 6 months
  The T score is a technical skills assessment score adapted to the scenarios of this study and based on the Formalized Recommendations of Experts published by the SFAR and the guidelines of the European Resuscitation Council
sense of self-efficacy (SEP) | 6 months
  To evaluate this SEP, we will use a visual analog scale: it will be represented by a horizontal line on which the participants will have to put a vertical line.
  This scale will be written out of 100, the score will be determined by the distance (in mm) that separates the left side of the horizontal line from the vertical line affixed by the participant. The leftmost part will correspond to 'I feel totally capable', the right part to 'I feel totally incapable'.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No